CLINICAL TRIAL: NCT06118307
Title: Shanghai Ovarian Cancer and Family Care Project
Status: Recruiting | Type: Observational
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS23259
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ambispective patient cohort: Patients attending the oncology department require differential diagnosis of ovarian cancer.
- High-risk population cohort: Family members of ovarian cancer patients; family history of BRCA mutation-related disease; abnormal findings on ovarian cancer screening; history of ovarian disease and other risk factors.
- Healthy control cohort: Healthy women with normal health examination results.

SUMMARY:
Ovarian cancer is the most lethal gynaecological malignancy, but its incidence in the general population is low. Due to the lack of effective prevention and successful screening approaches, most cases are diagnosed at advanced stages, leading to poor prognosis. In order to address the research requirements pertaining to ovarian cancer, the Shanghai Ovarian Cancer and Family Care Project was established. This initiative offers hospital-based resources for investigating ovarian cancer and high-risk populations. The project comprises an on-going ovarian cancer cohort, a high-risk population cohort, and a healthy population cohort. By leveraging these comprehensive cohorts, the project provides a unique platform for in-depth studies on the detection, prevention, early diagnosis, treatment, and prognosis of ovarian cancer.

ELIGIBILITY:
Participant meet the criteria for one of the following conditions:

* Patients attending the oncology department require differential diagnosis of ovarian cancer.
* Patients with known high-risk factors for ovarian cancer, such as history of ovarian cancer or BRCA-associated cancer, etc.
* Patients attending the Physical Examination Center who have normal findings on physical examination and no symptoms.

Exclusion Criteria:

* Individuals with evidence of another active cancer.
* Individuals who have prior bilateral oophorectomy.
* Individuals who are unwilling or unable to sign the informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the oncology department; patients with known risk factors for ovarian cancer; healthy individuals who are in good health determined by physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 3546 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2028-10-13 (Estimated); Study Completion 2028-10-13 (Estimated)

PRIMARY OUTCOMES:
Death due to ovarian cancer | From diagnosis of ovarian cancer until October 31, 2028.
  Death due to ovarian cancer determined by independent outcomes committee.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first maternity and infant hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Shi W, Zhang Y, Cheng S, Zhao Y, Li N, Li Y, Yang Y, Ding H, Li Z, Wang Y. Protocol of the SOCFC project: a longitudinal cohort study of ovarian cancer patients, high-risk populations, and healthy controls to identify factors and biomarkers associated with disease diagnosis and prognosis. BMC Cancer. 2025 Feb 26;25(1):355. doi: 10.1186/s12885-025-13652-9. PMID 40012035